CLINICAL TRIAL: NCT01551459
Title: A Randomised Phase II Study of Sunitinib Versus Dacarbazine in the Treatment of Patients With Metastatic Uveal Melanoma
Brief Title: A Phase II Study of Sunitinib Versus Dacarbazine in the Treatment of Patients With Metastatic Uveal Melanoma
Acronym: SUAVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Clatterbridge Cancer Centre NHS Foundation Trust (Other)
Collaborators: Cancer Research UK (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2008-008794-55; 2008-008794-55 (EudraCT Number); 8440 (Other: UKCRN); 75033520 (Other: ISRCTN); 10/H0904/15 (Other: Sunderland Research Ethics Committee)
Record Dates: First submitted 2012-03-08; First posted 2012-03-12 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2019-05

CONDITIONS: Metastatic Uveal Melanoma
Keywords: Uveal; Melanoma; Metastatic; Sunitinib
MeSH Terms: conditions — Uveal Melanoma; Melanoma; Neoplasm Metastasis | interventions — Dacarbazine; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Dacarbazine (Active Comparator): Patients will receive 1000mg/m2 every 21 days by IV until progression or unacceptable toxicity.
  Interventions: Drug: Dacarbazine
- Arm 2: Sunitinib (Experimental): Sunitinib: Patients will take 50mg orally once a day, for 28 days followed by a 14 day break, until progression or unacceptable toxicity.
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Dacarbazine — Dacarbazine: Patients will receive 1000mg/m2 every 21 days by IV until progression or unacceptable toxicity.
  Other Names: DTIC
  Arms: Arm 1: Dacarbazine
Drug: Sunitinib — Sunitinib: Patients will take 50mg orally once a day, for 28 days followed by a 14 day break, until progression or unacceptable toxicity
  Other Names: Sutent; Sunitinib Malate
  Arms: Arm 2: Sunitinib

SUMMARY:
Doctors usually treat uveal melanoma with radiotherapy or surgery. But if this cancer spreads, it is more difficult to treat.

Doctors usually treat uveal melanoma that has spread with a chemotherapy called dacarbazine, but they are always looking to find new ways to treat uveal melanoma.

This study aims to find out how well Sunitinib works to treat uveal melanoma and to see how long Sunitinib and Dacarbazine can help to prevent the cancer from getting worse.

DETAILED DESCRIPTION:
124 eligible patients will be randomised to either Sunitinib or Dacarbazine treatment. Participants will then attend 3-weekly clinic visits and undergo 12-weekly tumour assessment (CT or MRI scan) until disease progression (according to RECIST 1.1) has been identified.

At progression, patients may crossover to the other study treatment and continue with 3-weekly clinic visits and 12-weekly imaging until second progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed unresectable, metastatic uveal melanoma (histology must be available from a metastatic site)
* Patients with disease that is not amenable to surgery, radiation, or combined modality therapy with curative intent No prior systemic therapy for advanced disease, including regional delivery of drug therapy (prior surgery or radiofrequency ablation is acceptable)
* Patients who have received prior radiotherapy are eligible, however, measurable lesions must not have been previously irradiated
* Life expectancy > 12 weeks ECOG Performance status 0, 1 or 2
* At least one measurable target lesion, for further evaluation according to the Response Evaluation Criteria In Solid Tumours - RECIST version 1.1 completed within 28 days of randomisation
* Aged > 18 years
* Adequate haematological, renal and liver function as defined below and performed within 14 days of study inclusion:

Hb > 10 g/dl, platelets > 100 x109/L, WCC > 3.0 x109/L, ANC > 1.5x109/L, Bili < 1.5 x ULN, Alk phos < 5 x ULN, transaminases < 5 x ULN, Cr < 1.5 x ULN

* Able to provide written informed consent
* Females of child-bearing potential who have a negative pregnancy test prior to study entry and be using adequate contraception, which they agree to continue for 12 months after the study treatment

Exclusion Criteria:

Patients who have:

* Conjunctival melanoma
* Received any previous systemic therapy for uveal melanoma
* Known leptomeningeal or brain metastases
* Patients with a history of prior malignant disease (unless they have had more than 3 years free of disease or have had adequately treated non-melanomatous skin cancer or in situ carcinoma of the cervix)
* Had treatment with potent CYP3A4 inhibitors and inducers within 7 and 12 days respectively, prior to study treatment administration
* Therapeutic anticoagulation for treatment of DVT/PE. Concomitant treatment with therapeutic doses of anticoagulants (low dose warfarin up to 2mg PO daily for deep vein thrombosis prophylaxis is allowed)
* Unstable systemic diseases including uncontrolled hypertension (>150/100 mmHg despite optimal medical therapy) or active uncontrolled infections
* Any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism
* Clinically significant abnormal cardiac function with abnormal 12 lead ECG. Ongoing cardiac dysrhythmias of NCI CTCAE grade 2, poorly controlled atrial fibrillation of any grade, or prolongation of the QTc interval to >450 msec for males or >470 msec for females
* Any other serious or uncontrolled illness which, in the opinion of the investigator, makes it undesirable for the patient to enter the trial
* Any medical or psychiatric condition which would influence the ability to provide informed consent
* Pregnant or lactating women Lack of informed consent
* Any previous investigational agent within the last 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2010-10; Primary Completion 2017-09 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | Once all patients have been followed up for at least 3 months
  The primary outcome measure for this trial is the progression-free survival time measured from date of randomisation. For patients with evidence of progressive disease (as measured by CT scan, or MRI if necessary) or patients who have died from any cause, progression-free survival time will be calculated to date of progressive disease or date of death (whichever occurs first) and will be counted as events in the analysis. Patients still alive with no evidence of progression at the time of their last visit are censored at the time of the most recent information.

SECONDARY OUTCOMES:
Overall Survival | Analysis will take place once all patients have been followed up for at least 3 months
  Overall survival will be measured from date of randomisation to the date of death from any cause. Patients still alive at the time of the analysis are censored at the date of the most recent follow-up.
Overall Response Rate | Analysis will take place once all patients have been followed up for at least 3 months
  Overall response rate is defined as the proportion of complete (CR) or partial responders (PR) as defined by the RECIST version 1.1
Time to progression on first-line treatment compared to second-line treatment | Analysis will take place once all patients have been followed up for at least 3 months
  Time to progression on first-line treatment compared to second-line treatment for patients who receive cross-over therapy.
Overall response rate on first-line treatment compared to overall response rate on second-line treatment for patients who receive cross-over therapy | Analysis will take place once all patients have been followed up for at least 3 months
  Overall response rate on first-line treatment compared to overall response rate on second-line treatment for patients who receive cross-over therapy
Assessment of Adverse Events | Analysis will take place once all patients have been followed up for at least 3 months
  Adverse Events recorded following randomisation will be classified using NCI CTCAE version 4.

CONTACTS AND LOCATIONS:
Overall Officials: Ernest Marshall, Principal Investigator — The Clatterbridge Cancer Centre NHS Foundation Trust
Locations (1):
- Clatterbridge Centre for Oncology NHS Foundation Trust, Metropolitan Borough of Wirral, United Kingdom

REFERENCES:
- See also: Related Info: Liverpool Cancer Trials Unit — http://www.lctu.org.uk
- See also: Related Info — http://cancerhelp.cancerresearchuk.org/trials/a-study-looking-possible-new-treatment-for-eye-cancer-uveal-melanoma-suave